CLINICAL TRIAL: NCT00568685
Title: A Phase 3b, Randomized, Open-Label Assessment of Response to Various Doses of Atomoxetine Hydrochloride in Korean Pediatric Outpatients With Attention-Deficit/Hyperactivity Disorder
Brief Title: Atomoxetine to Treat Korean Children and Adolescents With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11710; B4Z-KL-LYEC
Record Dates: First submitted 2007-12-04; First posted 2007-12-06 (Estimated); Results first posted 2009-12-14 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atomoxetine 0.2 milligram per kilogram per day (mg/kg/day) (Active Comparator)
  Interventions: Drug: Atomoxetine Hydrochloride
- Atomoxetine 0.5 mg/kg/day (Active Comparator)
  Interventions: Drug: Atomoxetine hydrochloride
- Atomoxetine 1.2 mg/kg/day (Active Comparator)
  Interventions: Drug: Atomoxetine hydrochloride

INTERVENTIONS:
Drug: Atomoxetine Hydrochloride — Patients receive 0.2 mg/kg/day atomoxetine administered orally in two divided doses for the duration of the 6-week acute treatment period
  Other Names: LY139603; Strattera
  Arms: Atomoxetine 0.2 milligram per kilogram per day (mg/kg/day)
Drug: Atomoxetine hydrochloride — Patients receive 0.5 mg/kg/day atomoxetine administered orally in two divided doses for the duration of the 6-week acute treatment period
  Other Names: LY139603; Strattera
  Arms: Atomoxetine 0.5 mg/kg/day
Drug: Atomoxetine hydrochloride — Patients initially receive atomoxetine 0.5 mg/kg/day administered orally in two divided doses for approximately 7 days. Patients will then receive atomoxetine 0.8 mg/kg/day administered orally in two divided doses for approximately 7 days.
  Patients will receive atomoxetine 1.2 mg/kg/day administered orally in two divided doses for the remainder of the study, lasting approximately 28 days
  Other Names: LY139603; Strattera
  Arms: Atomoxetine 1.2 mg/kg/day

SUMMARY:
The purpose of this study is to provide information regarding the relative effectiveness of three different atomoxetine doses in the treatment of Korean children and adolescents with Attention-Deficit/Hyperactivity Disorder (ADHD)

ELIGIBILITY:
Inclusion Criteria:

* Patients will be outpatients who are aged 6 to 18 years old at the initial screening visit.
* Patients must have ADHD, based on the accepted criteria for that disease
* Patients must not have taken any medication used to treat ADHD for at least two weeks prior to beginning study treatment; and at least one week prior to the study screening visit during which initial ADHD assessments were made
* Patients must be able to swallow capsules
* Patients and parents (or legal guardians) must be judged by the study investigator to be reliable to keep appointments for clinic visits and all tests, including blood tests and any other required examinations

Exclusion Criteria:

* Patients must not have received any treatment within the last 30 days with a drug that has not been approved by their country's appropriate government agency
* Patients will not be included in the study if they have previously experienced any unwanted effects or serious medical events during atomoxetine treatment
* Patients will not be included in the study if they are judged by the study investigator to be at serious suicidal risk
* Patients will not be included in the study if they have cardiovascular disease or other conditions that could be worsened by an increased heart rate or increased blood pressure

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 153 (Actual)
Dates: Start 2007-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- South Korea (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine 0.2 Milligrams Per Kilogram, Per Day (mg/kg/Day): Patients receive 0.2 mg/kg/day atomoxetine administered orally in two divided doses for the duration of the 6-week acute treatment period.
- Atomoxetine 0.5 mg/kg/Day: Patients receive 0.5 mg/kg/day atomoxetine administered orally in two divided doses for the duration of the 6-week acute treatment period.
- Atomoxetine 1.2 mg/kg/Day: Patients initially receive atomoxetine 0.5 mg/kg/day administered orally in two divided doses for approximately 7 days. Patients will then receive atomoxetine 0.8 mg/kg/day administered orally in two divided doses for approximately 7 days. Patients will receive atomoxetine 1.2 mg/kg/day administered orally in two divided doses for the remainder of the study, lasting approximately 28 days.
Period: Overall Study
Arm/Group | Atomoxetine 0.2 Milligrams Per Kilogram, Per Day (mg/kg/Day) | Atomoxetine 0.5 mg/kg/Day | Atomoxetine 1.2 mg/kg/Day
Started | 51 | 51 | 51
Completed | 41 | 46 | 46
Not Completed | 10 | 5 | 5
Not completed — Adverse Event | 2 | 3 | 3
Not completed — Withdrawal by Subject | 7 | 2 | 2
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine 0.2 mg/kg/Day: Patients receive 0.2 mg/kg/day atomoxetine administered orally in two divided doses for the duration of the 6-week acute treatment period.
- Total: Total of all reporting groups
Arm/Group | Atomoxetine 0.2 mg/kg/Day | Atomoxetine 0.5 mg/kg/Day | Atomoxetine 1.2 mg/kg/Day | Total
Number analyzed (Participants) | 51 | 51 | 51 | 153
Age Continuous [Median (Inter-Quartile Range); unit: years] | 8.87 (2.774) [7.63 to 12.09] | 10.06 (2.178) [8.11 to 11.17] | 9.29 (2.187) [8.02 to 11.06] | 9.41 (2.382) [7.87 to 11.22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 41 | 40 | 85
  Male | 47 | 10 | 11 | 68
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 51 | 51 | 51 | 153
Age-Categorical [Number; unit: participants] — Pediatric participant age categories
  participants
    6-12 years | 38 | 44 | 44 | 126
    13-18 years | 13 | 7 | 7 | 27
Race/Ethnicity [Number; unit: participants]
  Korean | 51 | 51 | 51 | 153
ADHD Rating Scale-IV-Parent:Investigator Rated Hyperactivity Subscale Score [Mean (Standard Deviation); unit: units on a scale] — Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered and Scored (ADHDRS-IV-Parent:Inv) is an 18-item scale with one item for each of 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnosis for ADHD. Hyperactive/Impulsive Subscale consists of 9 items. Each item is scored on a 4 point scale (0=never or rarely; 1=sometimes; 2=often; 3=very often) for total score range of 0 (no symptoms) to 27 (highly symptomatic).
  units on a scale | 17.51 (5.825) | 16.61 (5.107) | 15.96 (5.553) | 16.69 (5.504)
ADHRS-IV-Parent: Inv. Inattention Subscale Score [Mean (Standard Deviation); unit: units on a scale] — Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered and Scored (ADHDRS-IV-Parent:Inv) is an 18-item scale with one item for each of 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnosis for ADHD. Inattention Subscale consists of 9 items. Each item is scored on a 4 point scale (0=never or rarely; 1=sometimes; 2=often; 3=very often) for total score range of 0 (no symptoms) to 27 (highly symptomatic).
  units on a scale | 21.57 (3.312) | 21.06 (3.630) | 20.20 (3.476) | 20.94 (3.499)
ADHRS-IV-Parent: Inv. Total Scores [Mean (Standard Deviation); unit: units on a scale] — Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered and Scored (ADHDRS-IV-Parent:Inv) is an 18-item scale with one item for each of 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) diagnosis for ADHD. Total Score consists of all 18 items. Each item is scored on a 4 point scale (0=never or rarely; 1=sometimes; 2=often; 3=very often) for total score range of 0 (no symptoms) to 54 (highly symptomatic).
  units on a scale | 39.08 (7.896) | 37.67 (7.064) | 36.16 (7.341) | 37.63 (7.489)
Clinical Global Impressions-Attention-Deficit/Hyperactivity Disorder Severity Scale (CGI-ADHD-S) [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impressions-Attention-Deficit/Hyperactivity Disorder Severity Scale (CGI-ADHD-S) rates severity using a 7-point scale (1=normal, not at all ill; 7=among the most extremely ill subjects). A higher score indicates greater severity of ADHD symptoms.
  units on a scale | 5.35 (0.688) | 5.31 (0.787) | 5.16 (0.703) | 5.27 (0.728)
Weight [Mean (Standard Deviation); unit: kilograms] | 35.67 (12.348) | 35.54 (10.647) | 35.48 (11.536) | 35.56 (11.455)

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Severity Scale (CGI-ADHD-S) Score at Days 7, 14, 42, and Last Observation Carried Forward Endpoint
Description: Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: Baseline, Days 7, 14, 42
Population: ITT population; last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine 0.2 mg/kg/Day | Atomoxetine 0.5 mg/kg/Day | Atomoxetine 1.2 mg/kg/Day
Number analyzed (Participants) | 51 | 51 | 51
units on a scale
  Day 7 | -0.24 (0.480) | -0.53 (0.612) | -0.30 (-.036)
  Day 14 | -0.73 (0.736) | -0.90 (0.918) | -0.92 (0.786)
  Day 42 | -1.04 (0.729) | -1.30 (1.121) | -1.56 (1.090)
  LOCF Endpoint | -0.98 (0.750) | -1.22 (1.119) | -1.54 (1.073)
Statistical Analysis 1: Comparison: Atomoxetine 0.2 mg/kg/Day vs Atomoxetine 0.5 mg/kg/Day vs Atomoxetine 1.2 mg/kg/Day; Test type: Superiority or Other; p = 0.0048, Mixed Models Analysis — This is the p value for CGI-ADHD-S score change at endpoint

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Improvement Scale (CGI-ADHD-I) Score at Days 7, 14, 42, and Last Observation Carried Forward Endpoint
Description: Measures total improvement (or worsening) of a patient's ADHD symptoms from the beginning of treatment. (1=very much improved, 7=very much worsened)
Time Frame: Baseline, Days 7, 14, 42
Population: ITT population; LOCF
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine 0.2 mg/kg/Day | Atomoxetine 0.5 mg/kg/Day | Atomoxetine 1.2 mg/kg/Day
Number analyzed (Participants) | 51 | 51 | 51
units on a scale
  Day 7 | 3.57 (0.645) | 3.22 (0.642) | 3.54 (0.813)
  Day 14 | 3.25 (0.729) | 3.20 (0.957) | 2.98 (0.721)
  Day 42 | 3.24 (0.970) | 3.09 (0.952) | 2.77 (0.973)
  LOCF Endpoint | 3.29 (0.957) | 3.16 (0.946) | 2.80 (0.969)
Statistical Analysis 1: Comparison: Atomoxetine 0.2 mg/kg/Day vs Atomoxetine 0.5 mg/kg/Day vs Atomoxetine 1.2 mg/kg/Day; Test type: Superiority or Other; p = 0.0153, Mixed Models Analysis — This is the p value for CGI-ADHD-I score change at endpoint

3. Secondary Outcome: Adverse Events Leading to Discontinuation
Description: Adverse Events (Preferred Term) leading to discontinuation by decreasing frequency
Time Frame: Baseline to Day 42
Population: As-treated population
Measure: Number; unit: events
Groups:
- 0-0.35 mg/kg/Day: Patients received atomoxetine 0-0.35 mg/kg/day
- 0.36-0.85 mg/kg/Day: Patients received atomoxetine 0.36-0.85 mg/kg/day
- > 0.85 mg/kg/Day: Patients received atomoxetine >0.85 mg/kg/day
Arm/Group | 0-0.35 mg/kg/Day | 0.36-0.85 mg/kg/Day | > 0.85 mg/kg/Day
Number analyzed (Participants) | 51 | 54 | 48
events
  Anorexia | 0 | 1 | 0
  Appendicitis | 0 | 1 | 0
  Dizziness | 0 | 1 | 0
  Dysphemia | 0 | 0 | 1
  Irritability | 1 | 0 | 0
  Sedation | 0 | 0 | 1
  Decreased appetite | 0 | 1 | 0
Statistical Analysis 1: Comparison: 0-0.35 mg/kg/Day vs 0.36-0.85 mg/kg/Day vs > 0.85 mg/kg/Day; Test type: Superiority or Other; p = .4500, Fisher Exact — P-value relates to the sum of adverse events leading to discontinuation

4. Primary Outcome: Change From Baseline to Day 42 Endpoint in Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version: Investigator Administered and Scored (ADHDRS-IV-Parent:Inv) Total Score
Description: Measures the 18 symptoms contained in the DSM-IV diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 none/never or rarely) to 3 (severe/very often). Total scores range from 0 (no symptoms) to 54 (highly symptomatic).
Time Frame: Baseline, Day 42
Population: Analysis included all randomized participants (intent-to-treat population)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Atomoxetine 0.2 mg/kg/Day | Atomoxetine 0.5 mg/kg/Day | Atomoxetine 1.2 mg/kg/Day
Number analyzed (Participants) | 51 | 51 | 51
units on a scale | -9.55 (7.758) [-12.03 to -7.07] | -12.31 (7.064) [-14.76 to -9.85] | -14.51 (7.216) [-16.99 to -12.04]
Statistical Analysis 1: Comparison: Atomoxetine 0.2 mg/kg/Day vs Atomoxetine 0.5 mg/kg/Day vs Atomoxetine 1.2 mg/kg/Day; Test type: Superiority or Other; p = 0.0240, ANCOVA

5. Secondary Outcome: Incidence of Completion of the Columbia Suicide-Severity Rating Scale, Suicide and Self-Harm Summary
Description: Columbia Suicide-Severity Rating Scale (C-SSRS) captures occurrence, severity & frequency of suicide-related thoughts & behaviors, via questions designed to solicit information to determine if a suicide-related thought or behavior occurred. The C-SSRS is not scored; recorded incidents are counted. C-SSRS was only required if an adverse event was reported that the investigator suspected to represent a suicidal thought or behavior. If the C-SSR was completed at a visit, the Self-Harm Supplement was also required. If a self-harm event was reported, the Self-Harm Follow-Up form was also required.
Time Frame: Baseline to Day 42
Population: As treated population
Measure: Number; unit: participants
Groups:
- >0.85 mg/kg/Day: Patients received atomoxetine >0.85 mg/kg/day
Arm/Group | 0-0.35 mg/kg/Day | 0.36-0.85 mg/kg/Day | >0.85 mg/kg/Day
Number analyzed (Participants) | 51 | 54 | 48
participants | 0 | 0 | 0

6. Secondary Outcome: Heart Rate Change From Baseline to Day 42 Endpoint
Time Frame: Baseline, Day 42
Population: ITT population
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Atomoxetine 0.2 mg/kg/Day | Atomoxetine 0.5 mg/kg/Day | Atomoxetine 1.2 mg/kg/Day
Number analyzed (Participants) | 51 | 51 | 51
beats per minute (bpm)
  Baseline | 87.86 (12.324) | 85.78 (10.769) | 90.10 (12.852)
  Day 42 | 90.43 (10.278) | 90.35 (11.028) | 93.89 (13.287)
  Change at endpoint | 2.59 (13.041) | 5.24 (13.621) | 4.98 (14.649)
Statistical Analysis 1: Comparison: Atomoxetine 0.2 mg/kg/Day vs Atomoxetine 0.5 mg/kg/Day vs Atomoxetine 1.2 mg/kg/Day; Test type: Superiority or Other; p = 0.8005, ANOVA — This is the p value for heart rate change at endpoint

7. Secondary Outcome: Temperature Change From Baseline to Day 42 Endpoint
Time Frame: Baseline, Day 42
Population: ITT population
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Atomoxetine 0.2 mg/kg/Day | Atomoxetine 0.5 mg/kg/Day | Atomoxetine 1.2 mg/kg/Day
Number analyzed (Participants) | 51 | 51 | 51
degrees Celsius
  Baseline | 36.63 (0.260) | 36.56 (0.397) | 36.50 (0.400)
  Day 42 | 36.58 (0.331) | 36.55 (0.332) | 36.59 (0.270)
  Change at endpoint | -0.05 (0.343) | -0.02 (0.339) | 0.07 (0.327)
Statistical Analysis 1: Comparison: Atomoxetine 0.2 mg/kg/Day vs Atomoxetine 0.5 mg/kg/Day vs Atomoxetine 1.2 mg/kg/Day; Test type: Superiority or Other; p = 0.4128, ANOVA — This is the p value for temperature change at endpoint

8. Secondary Outcome: Blood Pressure Change From Baseline to Day 42 Endpoint
Time Frame: Baseline, Day 42
Population: ITT population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Atomoxetine 0.2 mg/kg/Day | Atomoxetine 0.5 mg/kg/Day | Atomoxetine 1.2 mg/kg/Day
Number analyzed (Participants) | 51 | 51 | 51
mmHg
  Systolic Baseline | 105.98 (12.888) | 102.49 (11.279) | 106.12 (13.749)
  Systolic Day 42 | 107.82 (14.440) | 104.98 (10.988) | 108.48 (11.067)
  Systolic Change at Endpoint | 0.98 (16.535) | 2.35 (12.122) | 1.72 (13.391)
  Diastolic Baseline | 66.53 (10.567) | 65.39 (11.742) | 66.78 (11.524)
  Diastolic Day 42 | 67.45 (10.199) | 68.78 (11.677) | 70.02 (8.734)
  Diastolic Change at Endpoint | 0.16 (13.201) | 3.65 (12.058) | 2.17 (13.200)
Statistical Analysis 1: Comparison: Atomoxetine 0.2 mg/kg/Day vs Atomoxetine 0.5 mg/kg/Day vs Atomoxetine 1.2 mg/kg/Day; Test type: Superiority or Other; p = 0.9761, ANOVA — This is the p value for systolic change at endpoint
Statistical Analysis 2: Comparison: Atomoxetine 0.2 mg/kg/Day vs Atomoxetine 0.5 mg/kg/Day vs Atomoxetine 1.2 mg/kg/Day; Test type: Superiority or Other; p = 0.6419, ANOVA — This is the p value for diastolic change at endpoint

9. Secondary Outcome: Weight Change From Baseline to Day 42 Endpoint
Time Frame: Baseline, Day 42
Population: ITT population
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Atomoxetine 0.2 mg/kg/Day | Atomoxetine 0.5 mg/kg/Day | Atomoxetine 1.2 mg/kg/Day
Number analyzed (Participants) | 51 | 51 | 51
kilograms (kg)
  Baseline | 35.67 (12.348) | 35.54 (10.647) | 35.48 (11.536)
  Day 42 | 36.10 (12.524) | 35.72 (11.305) | 36.39 (11.708)
  Change at Endpoint | 0.37 (1.500) | -0.08 (1.155) | -0.15 (1.093)
Statistical Analysis 1: Comparison: Atomoxetine 0.2 mg/kg/Day vs Atomoxetine 0.5 mg/kg/Day vs Atomoxetine 1.2 mg/kg/Day; Test type: Superiority or Other; p = 0.2213, ANOVA — This is the p value for weight change at endpoint

ADVERSE EVENTS:
Description: The participant flow module encompasses the 'intention-to-treat' population. All safety data is reported with 'as-treated' population.
Groups:
- Atomoxetine 0.00-0.35 mg/kg/Day; Atomoxetine 0.36-0.85 mg/kg/Day; Atomoxetine >0.85 mg/kg/Day: Patients who received the actual dose range listed.
Arm/Group | Atomoxetine 0.00-0.35 mg/kg/Day | Atomoxetine 0.36-0.85 mg/kg/Day | Atomoxetine >0.85 mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 0/51 | 1/54 | 1/48
Other Adverse Events (participants affected / at risk) | 15/51 | 22/54 | 27/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine 0.00-0.35 mg/kg/Day (N=51) | Atomoxetine 0.36-0.85 mg/kg/Day (N=54) | Atomoxetine >0.85 mg/kg/Day (N=48)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine 0.00-0.35 mg/kg/Day (N=51) | Atomoxetine 0.36-0.85 mg/kg/Day (N=54) | Atomoxetine >0.85 mg/kg/Day (N=48)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 5 (5) | 4 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2)
Irritability (General disorders) | 2 (2) | 2 (2) | 4 (5)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 6 (8)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 4 (4)
Sleep disorder (Psychiatric disorders) | 4 (4) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days